CLINICAL TRIAL: NCT06113484
Title: Impact of a Mediterranean Diet (gReenheArTediEt - RATE) on Cardiovascular Disease Risk Factors: a Randomized Clinical Trial.
Brief Title: Impact of a Mediterranean Diet on Cardiovascular Disease Risk Factors
Acronym: RATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Católica Portuguesa (Other)
Collaborators: Associação para o Desenvolvimento do Centro Académico de Investigação e Formação Biomédica do Algarv (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22/2023/CEFCM
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Disease Risk
Keywords: Cardiovascular disease; Risk factors; Mediterranean Diet; Plant-based Diet
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DIET + EXERCISE (Experimental): This group engages in physical exercise plus a nutritional intervention. Monthly individual nutrition consultations are conducted. Additionally, this group also benefits from a group culinary workshop.
  Interventions: Other: DIET + EXERCISE
- WITHOUT DIET + EXERCISE (Other): This group engages in physical exercise; however, it is not the target of the nutritional intervention. Only a group educational session is conducted.
  Interventions: Other: WITHOUT DIET + EXERCISE
- WITHOUT DIET + WHITOUT EXERCISE (CONTROL) (No Intervention): This group does not engage in physical exercise, nor is it the target of the nutritional intervention. Only a group educational session is conducted.

INTERVENTIONS:
Other: DIET + EXERCISE — At first, a two-hour group session titled 'Discovering New Flavors' is conducted. This session aims to promote the consumption of healthy foods that should be included in the participants' daily diet. In order to create a different dynamic and enhance interaction, some recipe suggestions are prepared in a group setting. The intervention group is advised to have three (breakfast, lunch, and dinner) to four (breakfast, lunch, afternoon snack, and dinner) daily meals. Participants are encouraged not to count calories, thus emphasizing the importance of moderation. Regarding the main meals, legumes are recommended as a protein source for dinner. On the other hand, for lunch, the protein component can include white meats, fish, or eggs. Red and/or processed meats are excluded in this intervention. Moreover, all participants in this group are encouraged to practice a nightly fasting period of at least 12 hours.
  Arms: DIET + EXERCISE
Other: WITHOUT DIET + EXERCISE — An educational session titled "Healthy Eating: Nutritional Recommendations for Individuals at Risk of Cardiovascular Disease" will be conducted in a group setting.
  The objective of this session is to raise awareness among participants about the importance of a healthy diet and lifestyle in the prevention of cardiovascular diseases.
  Arms: WITHOUT DIET + EXERCISE

SUMMARY:
This approved and funded research project is part of a larger project titled "Algarve Active Ageing - Cardiac and Osteoarthritis Rehabilitation (A3-COR): personalized exercise protocol in the rehabilitation after acute myocardial infarction or at risk of cardiovascular disease and knee osteoarthritis, a multicenter clinical intervention study".

The main objective of this work is to quantify the effect of a nutritional and physical activity intervention in improving important risk factors for cardiovascular disease, such as body weight, body composition, and waist circumference.

DETAILED DESCRIPTION:
Cardiovascular diseases are the leading cause of death worldwide and one of the main contributors to diminished quality of life. It is estimated that in the year 2019, approximately 17.9 million individuals died due to this non-communicable disease, accounting for 32% of all global deaths. It is considered that CVDs result from the interaction between genetic predisposition (non-modifiable risk factors) and environmental influences (modifiable risk factors). Environmental factors prevail over others and often lead to negative outcomes through the adoption of poor lifestyles, such as imbalanced nutrition, physical inactivity, smoking, and alcohol habits. These are considered risk factors with direct effects on the pathogenesis of CVDs, and indirectly contribute to increasing the risk for predisposition to chronic diseases such as hypertension, dyslipidemia, overweight, obesity, and diabetes mellitus.

Currently, scientific literature has demonstrated the importance of diet in preventing CVDs and how it can minimize their risk factors. The Dietary Approaches to Stop Hypertension, Mediterranean dietary pattern, vegetarian diet, EAT-Lancet diet, and other dietary strategies have been published in various scientific journals.

Parallel to health, another topic that has gained prominence in the scientific community is environmental degradation derived from current food production. With the projected population growth until 2050, reaching 10 billion, the effects of food production on greenhouse gas emissions, nitrogen and phosphorus pollution, biodiversity loss, and water and land use are predicted to reach such high values that they will lead to the destabilization of the Earth system.

Considering that diet holds both environmental value and promotes cardiovascular health, this study aims to explore more sustainable and health-promoting dietary adaptations. This intervention will be based on principles of the Mediterranean diet, integrating higher consumption of plant sources compared to other mentioned patterns, and also leveraging the benefits of chronobiology, which are important for weight and adiposity control.

RECRUITMENT PLAN Participants will be recruited from the Algarve Active Ageing - Cardiac and Osteoarthritis Rehabilitation (A3-COR) project, carried out under the Algarve Biomedical Center - Research Institute. After the participants are integrated into the A3-COR project, those who meet the requirement of never having suffered from AMI but have high cardiovascular disease risk criteria according to the SCORE2 or SCORE2 O.P. algorithm will be contacted by phone. At this point, the objective of the nutritional intervention and the necessary conditions for participation will be explained (assessment of the remaining inclusion and exclusion criteria). After verifying these criteria, they will be invited to voluntarily participate in the present study. Those who accept to join the study will be contacted again to schedule the initial evaluation, and must sign the informed consent form prior to that.

PARTICIPANTS ALLOCATION Participants of the A3-COR control group who agree to participate in the present study (RATE) undergo an initial evaluation, forming the group (NO DIET + NO EXERCISE). These participants were randomly selected using new computer-generated numbers until a sample of 30-35 participants was reached from the total of 74 participants in this group. Participants from the Exercise Group of the A3-COR project who express interest in participating in the RATE project undergo randomization by numbers into one of two groups: the (EXERCISE + NO DIET n=30-35) group, which continues the exercise sessions as planned in the A3-COR project, and the (EXERCISE + DIET n=30-35) group, which, in addition to the exercise sessions, also receives nutritional guidance. This randomization is conducted among the 74 participants in the Exercise Group of the A3-COR project.

STATISTICS The statistical analysis will be performed using the Statistical Package for the Social Sciences (SPSS), version 27.0. All normally distributed numerical variables will be presented in the format of mean ± standard deviation. The normality of the variables will be tested using the Kolmogorov-Smirnov test. Differences between groups will be determined using paired t-tests. Repeated measures ANOVA will be used to detect changes between and within groups. Results will be considered statistically significant for p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 50 years
* Individuals meeting the criteria for high cardiovascular disease risk in the SCORE2 or SCORE2 O.P algorithm
* Autonomy in activities of daily living
* Provide informed and clarified consent

Exclusion Criteria:

* Occurrence of Acute Myocardial Infarction (AMI)
* To receive nutritional counseling from a registered dietitian
* To follow a vegetarian or strict vegetarian dietary pattern
* To take nutritional supplementation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-12-29 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Body weight (kg) | Day 1
  Medical Body Composition Analyzer - SECA® mBCA 514/515 - The subjects are placed standing on the scale in accordance with the manufacturer's instructions
Body weight (kg) | Day 90
  Medical Body Composition Analyzer - SECA® mBCA 514/515 - The subjects are placed standing on the scale in accordance with the manufacturer's instructions
Body fat (%) | Day 1
  Medical Body Composition Analyzer - SECA® mBCA 514/515 - The subjects are placed standing on the scale in accordance with the manufacturer's instructions.
Body fat (%) | Day 90
  Medical Body Composition Analyzer - SECA® mBCA 514/515 - The subjects are placed standing on the scale in accordance with the manufacturer's instructions.
Waist circumference (cm) | Day 1
  The abdominal circumference is assessed using a measuring tape at the midpoint between the upper edge of the iliac crest and the last palpable rib, following the methodology established by ISAK (International Society for the Advancement of Kinanthropometry)
Waist circumference (cm) | Day 90
  The abdominal circumference is assessed using a measuring tape at the midpoint between the upper edge of the iliac crest and the last palpable rib, following the methodology established by ISAK (International Society for the Advancement of Kinanthropometry)

SECONDARY OUTCOMES:
Lipid profile | Day 1
  Collection of a capillary blood sample by pricking the finger using a simple lancet. The COBAS b 101 system is used for evaluating the sample. The values presented refer to total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides.
Lipid profile | Day 90
  Collection of a capillary blood sample by pricking the finger using a simple lancet. The COBAS b 101 system is used for evaluating the sample. The values presented refer to total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides.
Hemoglobin A1c | Day 1
  Collection of a capillary blood sample by pricking the finger using a simple lancet. The COBAS b 101 system is used for evaluating the sample.
Hemoglobin A1c | Day 90
  Collection of a capillary blood sample by pricking the finger using a simple lancet. The COBAS b 101 system is used for evaluating the sample.
C-reactive protein | Day 1
  Collection of a capillary blood sample by pricking the finger using a simple lancet. The COBAS b 101 system is used for evaluating the sample.
C-reactive protein | Day 90
  Collection of a capillary blood sample by pricking the finger using a simple lancet. The COBAS b 101 system is used for evaluating the sample.
Hand grip strength | Day 1
  Measurement with the Lafayette Digital Hand Dynamometer 5030D1 on the dominant limb. The participant is seated with the elbow flexed at 90 degrees, the shoulder at 0 degrees of flexion, and the wrist in a neutral position. Three grips are performed with 30 seconds of rest between each, and the best of the three measurements is recorded.
Hand grip strength | Day 90
  Measurement with the Lafayette Digital Hand Dynamometer 5030D1 on the dominant limb. The participant is seated with the elbow flexed at 90 degrees, the shoulder at 0 degrees of flexion, and the wrist in a neutral position. Three grips are performed with 30 seconds of rest between each, and the best of the three measurements is recorded.
Sarcopenia | Day 1
  The SARC-F questionnaire, validated for the Portuguese population, is used for assessment.
  SARC-F scale scores range from 0 to 10 (i.e. 0-2 points for each component; 0 = best to 10 = worst) and were dichotomized to represent symptomatic (4+) vs. healthy (0-3) status.
Sarcopenia | Day 90
  The SARC-F questionnaire, validated for the Portuguese population, is used for assessment.
  SARC-F scale scores range from 0 to 10 (i.e. 0-2 points for each component; 0 = best to 10 = worst) and were dichotomized to represent symptomatic (4+) vs. healthy (0-3) status.
Fragility | Day 1
  The FRAIL Scale questionnaire, validated for the Portuguese population is used for assessment. The FRAIL scale includes 5 components: Fatigue, Resistance, Ambulation, Illness, and Loss of weight. Frail scale scores range from 0-5 (i.e., 1 point for each component; 0=best to 5=worst) and represent frail (3-5), pre-frail (1-2), and robust (0) health status.
Fragility | Day 90
  The FRAIL Scale questionnaire, validated for the Portuguese population is used for assessment. The FRAIL scale includes 5 components: Fatigue, Resistance, Ambulation, Illness, and Loss of weight. Frail scale scores range from 0-5 (i.e., 1 point for each component; 0=best to 5=worst) and represent frail (3-5), pre-frail (1-2), and robust (0) health status.
Food diary | Day 1
  The participants are asked to keep a three-day non-consecutive food diary (two weekdays and one weekend day) before and after the intervention.
Food diary | Day 90
  The participants are asked to keep a three-day non-consecutive food diary (two weekdays and one weekend day) before and after the intervention.
Cardiovascular Risk | Day 1
  The SCORE (Systematic COronary Risk Evaluation) algorithm is applied to individuals between the ages of 40 and 69.The SCORE2 algorithm is used in individuals aged between 70 and 89 years.
Cardiovascular Risk | Day 90
  The SCORE (Systematic COronary Risk Evaluation) algorithm is applied to individuals between the ages of 40 and 69.The SCORE2 algorithm is used in individuals aged between 70 and 89 years.
Bicep Skinfold | Day 1
  The measurement of bicep skinfold thickness is assessed according to the methodology established by ISAK (International Society for the Advancement of Kinanthropometry).
Bicep Skinfold | Day 90
  The measurement of bicep skinfold thickness is assessed according to the methodology established by ISAK (International Society for the Advancement of Kinanthropometry).
Tricep Skinfold | Day 1
  The measurement of tricep skinfold thickness is assessed according to the methodology established by ISAK (International Society for the Advancement of Kinanthropometry).
Tricep Skinfold | Day 90
  The measurement of tricep skinfold thickness is assessed according to the methodology established by ISAK (International Society for the Advancement of Kinanthropometry).
Arm circumference | Day 1
  The measurement of arm circumference is assessed according to the methodology established by ISAK (International Society for the Advancement of Kinanthropometry).
Arm circumference | Day 90
  The measurement of arm circumference is assessed according to the methodology established by ISAK (International Society for the Advancement of Kinanthropometry).
Lean body mass | Day 1
  Medical Body Composition Analyzer - SECA® mBCA 514/515 - The subjects are placed standing on the scale in accordance with the manufacturer's instructions.
Lean body mass | Day 90
  Medical Body Composition Analyzer - SECA® mBCA 514/515 - The subjects are placed standing on the scale in accordance with the manufacturer's instructions.
Arm muscle area | Day 1
  The formula suggested by Frisancho was used.
Arm muscle area | Day 90
  The formula suggested by Frisancho was used.
Legume intake | Day 1
  Number of plant-based meals (with legumes) per week.
Legume intake | Day 90
  Number of plant-based meals (with legumes) per week.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Católica Portuguesa, Porto, Portugal

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT06113484/Prot_SAP_ICF_000.pdf